CLINICAL TRIAL: NCT03182023
Title: Outcomes and Long-term Quality-of-life of Patients Treated With Extracorporeal Membrane Oxygenation
Brief Title: Long-term Outcome of Patients Treated With Extracorporeal Membrane Oxygenation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Dr., Southeast University, China
Other Study IDs: 20170606
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Long-term Outcome; Extracorporeal Membrane Oxygenation
Keywords: outcome,ECMO,Respiratory Failure,Circulatory Failure
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ECMO mode: ECMO mode includes Venovenous- ECMO and Venoarterial- ECMO

SUMMARY:
Outcomes and Long-term Quality-of-life of Patients Treated With Extracorporeal Membrane Oxygenation are not known in china.A cross-section survey will be performed to assess the long-term outcome of these patients.

DETAILED DESCRIPTION:
Patients admitted to ICUs and treated with extracorporeal membrane oxygenation from March 1,2011 to March 1,2017 were screened . Pre-Ecmo clinical parameters(diagnose,APACHE-II, SOFA,indications,expected mortality) and related treatment conditions(duration of ICU stay, duration of ECMO,duration of mechanical ventilation,ventilation conditions,prone ventilation,ECMO complications )will be used to assess the severity and curative effect of these patients.Short Form-36 Health Status Questionnaire,EuroQol-5 Dimensions and St. George's Respiratory Questionnaire(SGRQ) will deliver in these survivors ,which are used to assess the physical and mental health ,as well as the social adaptation. Finally a comprehensive assessment will be obtained to describe the outcomes and long-term quality-of-life of patients treated With ECMO.

ELIGIBILITY:
Inclusion Criteria:

* patients treated with ECMO

Exclusion Criteria:

* non-survivors of patients treated with ECMO，declined or lost to follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients treated with ECMO from January 1，2015 to March 1,2017
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Short Form-36 Health Status Questionnaire | June,2017-May,2018
  SF-36 is now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients.

SECONDARY OUTCOMES:
EuroQol-5 Dimensions | June,2017-May,2018
  The health-related quality of patients' life was rated with use of the EQ-5D index
the St. George's Respiratory Questionnaire(SGRQ) | June,2017-May,2018
  a fixed-format self-complete questionnaire for measuring health in chronic airflow limitation.Three component scores were calculated: symptoms, activity, and impacts (on daily life), and a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, Study Director — professor
Locations (1):
- Nanjing Zhong-Da Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No